CLINICAL TRIAL: NCT01787825
Title: Comparison of Capso Vision SV-1 to PillCam SB2 in the Evaluation of Subjects With Suspected Small Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capso Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Capso Vision SV-1
Record Dates: First submitted 2012-05-02; First posted 2013-02-11 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Intestinal Disease; Inflammatory Bowel Disease; Crohn Disease; Ulcer; Celiac Disease
Keywords: intestinal disease; inflammatory bowel disease; crohn disease; ulcer; celiac disease; angioectasia; polyp
MeSH Terms: conditions — Intestinal Diseases; Inflammatory Bowel Diseases; Crohn Disease; Ulcer; Celiac Disease; Polyps | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PillCam SB2 then CapsoCam SV-1 (Other): PillCam SB2 capsule then CapsoCam SV-1 capsule
  Interventions: Device: PillCam SB2 capsule; Device: CapsoCam SV-1
- CapsoCam SV-1 then PillCam SB2 (Other): CapsoCam SV-1 capsule then PillCam SB2 capsule
  Interventions: Device: PillCam SB2 capsule; Device: CapsoCam SV-1

INTERVENTIONS:
Device: PillCam SB2 capsule — Capsule Endoscopy system
  Other Names: capsule endoscopy system
Device: CapsoCam SV-1 — Capsule endoscopy
  Other Names: Capsule endoscopy

SUMMARY:
The purpose of this study is to compare the clinical findings involving the small bowel obtained with the Capso Vision Video Capsule Device to those results obtained with the PillCam SB2.

DETAILED DESCRIPTION:
This is a prospective, randomized, comparative multi-center site study. The study will be conducted at 5 to 10 clinical sites. Up to 120 subjects will be enrolled in the study in order to obtain complete endoscopic results involving at least 98 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 to 85 years of age (inclusive).
2. Willing and able to provide written informed consent.
3. Subjects with suspected small bowel disease who are referred for capsule endoscopy. Suspected small bowel disease includes suspected small bowel bleeding (including obscure gastrointestinal bleed), suspected or established Crohn's Disease [should have had patency capsule, CT or MR enterography before entry], suspected or known celiac disease, suspected small bowel tumor or familial polyposis syndrome.
4. If subject was referred for capsule endoscopy (CE) for identification of occult GI bleeding, has the subject undergone a non-diagnostic esophagoduodenoscopy and colonoscopy as part of their evaluation, OR has the subject had continued bleeding requiring transfusion since the initial evaluation, OR does the subject have the following hematocrit values <31% in males or <28% in females.

Exclusion Criteria:

1. Subjects who had a prior negative capsule endoscopy (within 1 year of study).
2. Known or suspected obstruction or stricture unless patency capsule confirms patency.
3. Known or suspected gastrointestinal perforation.
4. Known or suspected small bowel diverticuli.
5. Known swallowing disorder or the inability or unwillingness to swallow pills.
6. Radiation or chemotherapy induced enteritis.
7. History of Zenker's or known duodenal or jejunal diverticula.
8. Isolated diarrhea or isolated abdominal pain without alarm signs or symptoms
9. Subjects who are high risk for undergoing surgical interventions (i.e., to CONFIDENTIAL CapsoVision Protocol SV-1 Revision: October 17, 2011 7 remove the capsule when capsule retention occurs).
10. Subjects with DNR/DNI "do not resuscitate/do not intubate" status.
11. Known or suspected gastrointestinal dysmotility.
12. Presence of cardiac pacemaker, implanted defibrillator or other electromedical implant.
13. History of skin reaction to adhesives.
14. Subjects who in the Investigator's opinion should not consume the 2L GoLytely and 10 mg bisacodyl study drugs, because it could pose a significant additional risk to the subject because of the subject's medical condition.
15. Subjects who are scheduled for an MRI within 30 days of the last study visit.
16. Pregnancy; females of childbearing potential must have a negative urine pregnancy test at screening.
17. Prisoners.
18. Mental and/or physical condition precluding compliance with the study and/or device instructions.
19. Participation in another clinical study within past 30 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-05; Primary Completion 2015-04 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shabana F Pasha, MD, Principal Investigator — Mayo Clinic
Locations (7):
- United States (6):
  - Shabana F. Pasha, MD, Scottsdale, Arizona
  - Gastro Health, Miami, Florida
  - University of Massachusetts, Worcester, Worcester, Massachusetts
  - Medical University of South Carolina, Charleston, South Carolina
  - Ziad Younes, MD, Germantown, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
- Pacific Gastroenterology Associates GI Research Institute, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from population of patients prescribed capsule endoscopy for OGIB
Groups:
- CapsoCam SV-1 Then PillCam SB2: Participants first received CapsoCam SV-1 then 30-60 minutes later received Pillcam SB2
- PillCam SB2 Then CapsoCam SV-1: Participants first received PillCam SB2 then 30-60 minutes later receive CapsoCam SV-1
Period: Overall Study
Arm/Group | CapsoCam SV-1 Then PillCam SB2 | PillCam SB2 Then CapsoCam SV-1
Started | 60 | 61
Completed (This was a paired study with crossover with randomization.) | 54 | 60
Not Completed | 6 | 1
Not completed — Subject Did Not Ingest Capsules | 1 | 0
Not completed — Data Not Analyzable | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: PillCam SB2 capsule and CapsoCam SV-1 capsule in random order, PillCam SB2 capsule: Capsule Endoscopy system, CapsoCam SV-1: Capsule endoscopy
  The analysis population consisted of subjects that swallowed the capsules.
Arm/Group | All Study Participants
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (15.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 91
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 104
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Canada | 40
  United States | 80

OUTCOME MEASURES:

1. Primary Outcome: Normal vs Abnormal, Overall Impression
Description: The review of images of suspected diseased small bowel to determine agreement among readers between the two image capture systems: CapsoCam SV-1 and PillCam SB2. The proportion of Normal vs Abnormal, Overall Impression based upon the result of 2 out of 3 data readers in agreement.
Time Frame: Study Completion
Population: Note: Each participant swallowed both Pill Cam and CapsoCam approximately 30-60 minutes apart. the order in which the cams were swalloed was randomized.
Measure: Number; unit: participants
Groups:
- CapsoCam SV-1; PillCam SB2: Each participation swallowed both PillCam SB2 and CapsoCam SV-1 30-60 minutes apart. The order in which the cams were swallowed was randomized.
Arm/Group | CapsoCam SV-1 | PillCam SB2
Number analyzed (Participants) | 114 | 114
participants
  Abnormal | 42 | 42
  Normal | 72 | 72
Statistical Analysis 1: Comparison: CapsoCam SV-1 vs PillCam SB2; There was a comparison between normal and abnormal images. And detailed analysis of abnormal images that were considered clinical significant; Test type: Non-Inferiority — This is McNemar design; p = 1.0000, McNemar — The blinded readers assessed concordance of normal versus abnormal and overall concordance of clinically significant abnormal images; percentage concordance = 77.19, 95% CI 2-sided [68.68 to 83.93] — Overall concordance of clinically significant abnormal images

2. Secondary Outcome: Comparison of SB Transit Times With CapsoCam SV-1 and PillCam SB2
Description: Total transit time, was determined the time the 1st Duodenal image to the 1st cecal or IC Valve image as determined by the readers.
Time Frame: Study Completion
Population: For CapsoCam SV-1 data was captured for 112 subjects total transit time. For PillCam SB2, data was captured for 110 subjects for total transit time.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CapsoCam SV-1 | PillCam SB2
Number analyzed (Participants) | 112 | 110
hours | 4.1 (1.85) | 3.6 (1.56)

3. Secondary Outcome: Comparison of Diagnostic Yield of CapsoCam SV-1 as Compared to PillCam SB2
Description: Comparison of Diagnostic Yield of CapsoCam SV-1 as compared to PillCam SB: Proportion of primary diagnostic yields based upon the result of 2 out of 3 readers in agreement or the consensus group result.
Time Frame: Study Completion
Measure: Number; unit: participants
Arm/Group | CapsoCam SV-1 | PillCam SB2
Number analyzed (Participants) | 114 | 114
participants
  Normal | 71 | 70
  Vascular | 24 | 21
  Mass/Polyp | 1 | 4
  Blood | 1 | 3
  Ulcerative | 15 | 14
  Other | 2 | 2
Statistical Analysis 1: Comparison: CapsoCam SV-1 vs PillCam SB2; Test type: Superiority or Other; p = 0.972, Bowkers; percentage concordance = 71.93, 95% CI 2-sided [63.07 to 79.36]

4. Secondary Outcome: Preference Between CapsoCam SV-1 and PillCam SB2
Description: Subject preference between CapsoCam SV-1 and PillCam SB2 based on pill preference questionnaire administered to subjects
Time Frame: Study Completion
Population: For CapsoCam SV-1 and PillCam SB2 preference data was captured for 113 subjects.
Measure: Number; unit: participants
Groups:
- CapsoCam SV-1 Preference: Subject preference for CapsoCam SV-1
- PillCam SB2: Subject preference for PillCam SB2
Arm/Group | CapsoCam SV-1 Preference | PillCam SB2
Number analyzed (Participants) | 113 | 113
participants | 89 | 24

ADVERSE EVENTS:
Time Frame: Within 30 days of Subjects' Swallowing of both cpasules: CapsoCam SV-1 and PillCam SB2
Groups:
- All Study Participants: PillCam SB Capsule and CapsoCam SV-1
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 2/120
Other Adverse Events (participants affected / at risk) | 12/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=120)
Capsule Endoscope Retention (Gastrointestinal disorders) | 2 (2) — Capsule Endoscopes (Both CapsoCam SV-1 and PillCam SB2) retained within the small bowel of each of two (2) enrolled subjects. Capsules were removed via surgical intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=120)
GI Tract discomfort or pain and nausea (Gastrointestinal disorders) | 6 (6) — GI Tract discomfort or pain and nausea attributed to bowel preparation for the procedures by study investigators
Malaise (Gastrointestinal disorders) | 1 (1) — Malaise in one (1) subject
Skin Irritation and Itchiness (Skin and subcutaneous tissue disorders) | 2 (2) — Skin Irritation and itchiness secondary to adhesive tape used to secure PillCam SB2 wireless receiver
Delayed Capsule Excretion (Gastrointestinal disorders) | 1 (1) — Delayed Capsule Excretion: Capsule s not retrieved and returned to investigator/research site for analysis
Right Kidney Pain (Renal and urinary disorders) | 1 (1) — Right Kidney Pain: Cause unknown
Migraine Headache (Nervous system disorders) | 1 (1) — Migraine Headache in one (1) subject

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No